CLINICAL TRIAL: NCT02120846
Title: Effects of Flywheel Resistance Training on Cognitive Function in Stroke Patients
Acronym: KAROL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Rodrigo Fernandez Gonzalo, Ph.D., Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Flywheel stroke; 1301 (Other Grant/Funding Number: Tesch-Övermo Stiftelsen)
Record Dates: First submitted 2014-04-16; First posted 2014-04-23 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Stroke
Keywords: Stroke; Flywheel resistance exercise; Muscle function; Cognitive function
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Flywheel leg-press resistance exercise (Experimental): Participants from the resistance exercise group will perform a 12-wk unilateral flywheel resistance training program with the paretic limb. Four sets of seven coupled concentric and eccentric actions will be completed in the leg press device using flywheel technology twice weekly. Power in each set and repetition will be measured. During all training sessions, subjects will receive visual real-time feedback of power and force produced during each concentric-eccentric action.
  Interventions: Other: Flywheel leg-press resistance exercise
- Control (No Intervention): Daily routines

INTERVENTIONS:
Other: Flywheel leg-press resistance exercise
  Other Names: Yo-Yo Techonlogy
  Arms: Flywheel leg-press resistance exercise

SUMMARY:
Forty patients will be assigned to either a training group (12 wk unilateral knee extension flywheel resistance exercise; 4 sets of 7 reps 2 days/week) or a control group. Patients will maintain daily routines and any prescribed rehabilitation program. Established methods to assess muscle and cognitive function will be employed before and after the intervention.

This project will disclose whether an exercise paradigm, known to improve muscle function and increase muscle volume in healthy populations, will induce similar adaptations in chronic stroke patients. More importantly, this study will elucidate if any impairment in cognitive function caused by stroke, can be reversed with this particular resistance exercise regimen.

The information gained from this project will have significant implications and aid in advancing rehabilitation programs and exercise prescriptions for men and women suffering from stroke. The overall objective of this research is to promote independence and hence quality of life in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Mild-moderate hemiparetic gait
* > 6 months post-stroke
* Able to perform flywheel leg-press exercise

Exclusion Criteria:

* Unstable angina
* Congestive heart failure
* Severe arterial disease
* Major depression
* Dementia
* Chronic pain
* Psychotic alterations

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Cognitive Function at 3 months | Baseline, Month 3
  Cognitive function will be assessed before and after the training period in all participants. In a 60-90 min session, with 10 min of rest is needed, validated tests will be used to evaluate different domains of cognitive function: Speed of information processing; Short- and long-term memory; Attention; Language; Learning; Delayed recall; Working memory; Inhibition; Visuo-motor scanning; Dual task attention; Quality of life.
Change from baseline in Functional Performance at 3 months | Baseline, Month 3
  Up-and-Go, Fast Gait Speed, Berg Balance Scale
Change from baseline in Muscle Function at 3 months | Baseline, Month 3
  Isometric and dynamic force, and peak power during flywheel leg-press exercise. Quadriceps muscle volume (MRI).

SECONDARY OUTCOMES:
Change from baseline in Spasticity at 3 months | Baseline, Month 3
  Modified Ashworth Scale

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Fernandez-Gonzalo, Ph.D., Principal Investigator — Karolinska Institutet
Locations (1):
- Hospital Universitari Parc Tauli, Sabadell, Barcelona, Spain

REFERENCES:
- [Derived] Fernandez-Gonzalo R, Fernandez-Gonzalo S, Turon M, Prieto C, Tesch PA, Garcia-Carreira Mdel C. Muscle, functional and cognitive adaptations after flywheel resistance training in stroke patients: a pilot randomized controlled trial. J Neuroeng Rehabil. 2016 Apr 6;13:37. doi: 10.1186/s12984-016-0144-7. PMID 27052303